CLINICAL TRIAL: NCT02994095
Title: A Pilot Study of a Community Health Agent-led Diabetes Self-Management Program Using Motivational Interviewing-based Approaches in a Public Primary Care Center in São Paulo, Brazil
Brief Title: A Pilot Study of a Community Health Agent-led Diabetes Self-Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mary Ellen Michele Heisler, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00073693
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Pilot Projects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single intervention arm (Experimental): Trained CHAs in Motivational Interviewing in pilot study
  Interventions: Behavioral: Pilot Study

INTERVENTIONS:
Behavioral: Pilot Study — Trained community health agents used Motivational Interviewing-based counseling and action planning in monthly home visits with adults with diabetes

SUMMARY:
This was a pilot study to assess the feasibility and acceptability of training Community Health Agents in Motivational Interviewing in real-life primary care centers.

DETAILED DESCRIPTION:
Rates of noncommunicable diseases (NCDs) such as type 2 diabetes are escalating in low and middle-income countries such as Brazil. Scalable primary care-based interventions are needed to improve self-management and clinical outcomes of adults with diabetes. This pilot study examines the feasibility, acceptability, and outcomes of training community health agents (CHAs) in Motivational Interviewing (MI)-based counseling for patients with poorly controlled diabetes in a primary care center in São Paulo, Brazil.

Nineteen salaried CHAs participated in 32 hours of training in MI and behavioral action planning. With support from booster training sessions, they used these skills in their regular monthly home visits over a 6 month period with 57 diabetes patients with baseline HbA1cs > 7.0%. The primary outcome was patients' reports of the quality of diabetes care as measured by the Portuguese version of the Patient Assessment of Chronic Illness Care (PACIC) scale. Secondary outcomes included changes in patients' reported diabetes self-management behaviors and in A1c, blood pressure, cholesterol and triglycerides. CHAs' fidelity to and experiences with the intervention were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with T2 diabetes who received care at the primary care center
* A1c>7.0% in prior six months

Exclusion Criteria:

* Age> 75
* being pregnant
* having terminal health condition or other conditions that would impede participation such as dementia and mental illness

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
PACIC score | Six months
  Quality of Diabetes Care Received

CONTACTS AND LOCATIONS:
Overall Officials: Michele Heisler, MD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: Yes
De-identified data set available on request.

REFERENCES:
- [Derived] do Valle Nascimento TM, Resnicow K, Nery M, Brentani A, Kaselitz E, Agrawal P, Mand S, Heisler M. A pilot study of a Community Health Agent-led type 2 diabetes self-management program using Motivational Interviewing-based approaches in a public primary care center in Sao Paulo, Brazil. BMC Health Serv Res. 2017 Jan 13;17(1):32. doi: 10.1186/s12913-016-1968-3. PMID 28086870